CLINICAL TRIAL: NCT04073927
Title: The Butyful Study. Effect of Butyrate on Inflammation and Albuminuria in Patients With Albuminuria, Type 1 Diabetes and Intestinal Inflammation A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Butyrate on Inflammation and Albuminuria in Patients With Albuminuria, Type 1 Diabetes and Intestinal Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Folkhälsan Researech Center (Other)
Responsible Party: Principal Investigator, Peter Rossing, Professor, MD, DMsc, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-18062027
Record Dates: First submitted 2019-08-16; First posted 2019-08-29 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 1; Albuminuria
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Albuminuria | interventions — Butyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium butyrate (Active Comparator): 3.6 g sodium butyrate. 6 capsules twice daily for 12 weeks.
  Interventions: Dietary Supplement: Sodium butyrate
- Placebo (Placebo Comparator): Placebo. 6 capsules twice daily for 12 weeks.
  Interventions: Dietary Supplement: Sodium butyrate

INTERVENTIONS:
Dietary Supplement: Sodium butyrate — Sodium butyrate Class: Fatty acids Ingredients (100 g): Na-butyrate (50 g), acylglycerol (mono- di, -triacylglycerol; 42 g), bee wax (5 g), sodium alginate E401 (2 g), emulsifier (0.5 g).
  The capsules contain granulated sodium butyrate and are coated with a sodium alginate membrane.

SUMMARY:
The objective is to assess the impact of 12 weeks supplement of sodium-butyrate twice daily or placebo on intestinal inflammation and albuminuria.

A randomized, placebo-controlled, double-blind, two-site trial including 48 patients with type 1 diabetes, albuminuria and intestinal inflammation. Participants will be randomized 1:1 to active treatment or placebo for a period of 12 weeks.

The primary endpoint is change from baseline to week 12 in intestinal inflammation, measured by fecal calprotectin.

DETAILED DESCRIPTION:
In patients with type 1 diabetes, increased intestinal inflammation, reduced gut barrier function and resulting influx of proinflammatory molecules have been described. This might contribute to systemic inflammation and the development of diabetic complications like nephropathy and ischemic heart disease. Interestingly, the gut microbiota is altered in persons with type 1 diabetes, who have less butyrate-producing bacteria. The short-chain fatty acid butyrate improves the intestinal barrier function, and the altered bacterial composition is hypothesized to play a role in the intestinal inflammation. Treatment with butyrate has improved metabolic, colonic and renal function in animal models of chronic kidney disease.

The aim of the study is to test whether orally ingested sodium butyrate can reduce intestinal inflammation in patients with type 1 diabetes and albuminuria in a randomized, placebo-controlled, double-blind, two-site trial.

Persons with type 1 diabetes and albuminuria are recruited from Steno Diabetes Center Copenhagen (SDCC) and Folkhälsan Research Center, FinnDiane, Helsinki, Finland and screened for intestinal inflammation. 48 participants with intestinal inflammation (fecal calprotectin ≥50 μg/g) are randomized to receive 3.6 g sodium butyrate or placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age with a diagnosis of type 1 diabetes (age at onset <40 years; permanent insulin treatment initiated within 1 year of diagnosis)
2. Albuminuria: UACR > 30 mg/g documented in medical history
3. Calprotectin quick-test result ≥ 50 μg/g (CalDetect 50/200, Preventis) between visit 1 and visit 2.
4. Able to understand the written patient information and give informed consent

Exclusion Criteria:

1. Known inflammatory bowel disease
2. IBD symptoms due to investigators opinion
3. Known celiac disease
4. Existing ostomy
5. Known rheumatic disorders treated with anti-inflammatory agents
6. Known hyperthyroidism or hypothyroidism Butyful Protocol - page 12 - Version 3, 25.02.2019
7. Active immunosuppressant therapy with systemic effect due to investigator's opinion
8. Current cancer treatment or within five years from baseline (except basal cell skin cancer or squamous cell skin cancer)
9. eGFR<15, dialysis or kidney transplantation
10. Diagnosis of non-diabetic CKD
11. Active antibiotic therapy until 30 days ahead of screening
12. Unable to participate in study procedures
13. Not able to assess calprotectin by quick test in two attempts
14. Any clinically significant disorder, except for conditions associated with type 1 DM history, which in the Investigators opinion could interfere with the results of the trial
15. Pregnancy or lactation
16. Participation in another intervention study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-08-05 (Estimated); Study Completion 2020-08-05 (Estimated)

PRIMARY OUTCOMES:
Intestinal inflammation | Baseline to week 12
  Change in concentration of fecal calprotectin determined by ELISA

SECONDARY OUTCOMES:
Fecal intestinal alkaline phosphatase (IAP) | Baseline to week 12
  Change in IAP activity in feces assessed by colorimetric assay
Short-chain fatty acids (SCFAs) | Baseline to week 12
  Change in acetate, propionate, butyrate and valerate concentration in feces measured by gas chromatography-mass spectrometry
Albuminuria | Baseline to week 12
  Change in urinary albumin-creatinine ratio (UACR)
Kidney function | Baseline to week 12
  Change in eGFR

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, Professor, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (2):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark
- Folkhälsan Research Center, FinnDiane, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No